CLINICAL TRIAL: NCT06226311
Title: Environmental Pollutants in Pregnancy - Exposure Assessment and Association With Early Childhood Development - IoMumNEXT
Brief Title: Environmental Pollutants in Pregnancy - IoMumNEXT
Acronym: IoMumNEXT
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Universidade do Porto (Other)
Collaborators: Centro Hospitalar De São João, E.P.E. (Other); Centro de Investigação em Tecnologias e Serviços de Saúde (Other); Rede de Investigação em Saúde (Other)
Responsible Party: Sponsor
Other Study IDs: IoMumNEXT
Record Dates: First submitted 2022-12-06; First posted 2024-01-26 (Actual); Last update posted 2024-01-26 (Actual); Status verified 2023-10

CONDITIONS: Early Childhood, Neurodevelopment; Early Childhood, Anthropometry
Keywords: Pregnancy; Childhood; Exposure; Environmental Pollutants; Anthropometry
MeSH Terms: interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Urine samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Children of IoMum pregnants cohort: IoMum participants without congenital malformations or gestational diabetes, with a singleton pregnancy with live birth, who provided contact and a T1 urine sample, will be invited to participate under signed informed consent.
  Interventions: Other: Data collection; Other: Diagnostic Test: Urinary

INTERVENTIONS:
Other: Data collection — Collection of sociodemographic, lifestyle and health data; Child anthropometry (weight, height and head circumference) at the ages of 3-4 and 5-6 years Child neurodevelopment scores at the ages of 3-4 and 5-6 years
Other: Diagnostic Test: Urinary — Trichloro-pyridinol (TCPy) and 3-phenoxybenzoic acid (3-PBA) Environemental oligoelements including Lithium (7Li), Arsenic (75As), Cadmium (111Cd), Lead (208Pb) and Mercury (80Hg)

SUMMARY:
Globally 12.6 million people, including 1.7 million children under the age of 5, die each year from environmental-related illnesses. Prenatal exposure to environmental chemical pollutants has been associated with perinatal mortality, prematurity, low birth weight, congenital malformations, neurobehavioral function disorder and metabolic disorders. This project aims: a) to evaluate exposure to environmental pollutants during pregnancy; and, b) to study the association of this exposure with anthropometry and neurodevelopment of the offspring, up to 6 years of age. This study will be based on a population of 1000 pregnant women whose recruitment has already started under the IoMum project (clinical trials #NCT04010708), previously approved by Ethics Commitee of Centro Hospitalar e Universitário São João/Faculdade de Medicina da Universidade do Porto (#292-17). Maternal urine samples collected in the 1st and 3rd trimesters of pregnancy will be used. Maternal urinary concentrations of toxic metals and pesticide metabolites will be determined and neurodevelopmental outcomes will be evaluated as well as anthropometric parameters of children from birth to 6 years of age. The results of this project will contribute to the characterization of the exposure of Portuguese pregnant women to environmental pollutants as well as to the knowledge on the association between isolated or cumulative exposure to these pollutants and the health of the offspring.

DETAILED DESCRIPTION:
IoMumNEXT is a prospective observational study which will take advantage of our previous IoMum project - monitoring of iodine status in Portuguese pregnant women: impact of supplementation (Clinical Trials record: NCT04010708), a prospective observational study that has set up a cohort of 1155 pregnant women, living in the Porto and Lisbon Metropolitan Areas.

In a subsample of 199 pregnant women of this IoMum@Porto cohort it was already possible to conclude that:

1. 19 and 32% of women had urinary levels (first trimester) of lead (208Pb) and arsenic (75As), respectively above the corresponding reference values (> 4 microg / L for Pb and> 35 microg / L for As).
2. Maternal urinary Pb levels (first trimester) revealed a positive association with birth weight and length.
3. Maternal urinary levels of As (first trimester) revealed a positive association with head circumference at birth.
4. In a subsample of 69 pregnant women, 52% showed urinary 3-Phenoxybenzoic acid (3-PBA) levels above the detection level.

In addition to Pb, As and 3-PBA, the maternal urinary concentrations of other pollutants such as the elements lithium (7Li), cadmium (111Cd) and mercury (80Hg), and the pesticide metabolite trichloro-pyridinol (TCPY) will be analyzed. The continuity of this work will allow an important scientific advance, regarding the association between exposure to environmental pollutants and the physical and neurobehavioral development of children.

This proposal is in line with goal 3 (Health and well-being) of the United Nations Agenda 2030.

The study population will be composed of the pregnant women from the IoMum cohort as well as by their children born from this cohort. Maternal urine samples collected in the first trimester (T1) and third trimesters (T2) of pregnancy will be used, as well as urine samples from children collected between 3 and 6 years of age. Sociodemographic, lifestyle, anthropometric and health data will continue to be collected between 3 and 4 years of age (T3) and between 5 and 6 years of age (T4). Additionally, neurodevelopment will be assessed by Vineland adaptative behaviour scale at T3 and T4.

ELIGIBILITY:
Inclusion Criteria:

* Have had single live birth
* Have provided contact and a urine sample T1
* Have provided consent to participate at T1
* Have provided consent to participate at T3

Exclusion Criteria:

Pregnancy complications

* Congenital malformations
* Gestational diabetes

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The study population will be based on the 1155 pregnant women from the IoMum cohort, who have already been recruited at the Centro Hospitalar Universitário de São João (CHUSJ) and at CUF Descobertas Hospital (CUFD), Lisbon, in the 1st trimester ultrasound scan, as well as by the children born in this cohort.
Sampling Method: Non-Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2024-09-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Anthropometric measurements of children - Weight | The information will be collected at baseline by telephone contact (3-4 years of age) with parents or legal representatives or by direct, in person, measurement (5-6 years of age)
  Information n the weight (in kilograms) of children aged between 3-4 and 5-6 years will be recorded
Anthropometric measurements of children - Height | The information will be at baseline collected by telephone contact (3-4 years of age) with parents or legal representatives or by direct, in person, measurement (5-6 years of age)
  Information on the height (in centimeters) of children aged between 3-4 and 5-6 years will be recorded
Neurodevelopment scores of children | At 3-4 and 5-6 years old of the children, parents will answer a questionnaire regarding daily living, social, communication and motor skills adjusetd to the specific age group, at baseline
  Communication, daily life activities, socialization and motor skills will be assessed using the Vineland Adaptive Behavior Scale
1st trimester maternal urinary concentrations of environmental pollutants | Between gestational weeks 10 and 13 plus 6 days (Timepoint 1)
  Median urinary concentations of 3-PBA, TCPY in micrograms per liter
1st trimester maternal urinary concentrations of oligoelements | Between gestational weeks 10 and 13 plus 6 days (Timepoint 1)
  Median urinary concentations of Pb, As, Cd, Li, Hg in micrograms per liter

SECONDARY OUTCOMES:
1st trimester maternal urinary concentration of iodine | Between gestational weeks 10 and 13 plus 6 days (Timepoint 1)
  Median urinary iodine concentrations at 1st trimester of gestation, in micrograms per liter
3rd trimester maternal urinary concentration of environmental pollutants | Between gestational weeks 37 and 40 plus 6 days (Timepoint 2)
  Median urinary concentations of 3-PBA, TCPY, in micrograms per liter
3rd trimester maternal urinary concentration of oligoelements | Between gestational weeks 37 and 40 plus 6 days (Timepoint 2)
  Median urinary concentations of oligoelements including Pb, As, Cd, Li, Hg, in micrograms per liter
Anthropometric measures of the children at birth, 1, 2 and 4 years - Weight | Birth, 1, 2 and 4 years of age (retrospectively collected at the same moment, during the first phone call)
  Weight information in grams or kilograms will be collected retrospectively from the clinical records or reported by the parents
Anthropometric measures of the children at birth, 1, 2 and 4 years - Height | Birth, 1, 2 and 4 years of age (retrospectively collected at the same moment, during the first phone call)
  Stature information in centimeters will be collected retrospectively from the clinical records or reported by the parents
Anthropometric measures of the children at birth, 1 and 2 years - Head circumference | Birth, 1 and 2 years of age (retrospectively collected at the same moment, during the first phone call)
  Head circumference in centimeters will be collected retrospectively from the clinical records or reported by the parents
Apgar index | Birth (retrospectively collected)
  Apgar index at 1, 5 and 10 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Elisa Keating, PhD, Principal Investigator — Universidade do Porto
Locations (1):
- Faculty of Medicine (FMUP), Porto, Portugal